CLINICAL TRIAL: NCT05210426
Title: The Effects of Pilates on Posture and Physical Fitness Parameters in 5-6 Years Old Children: a Non-randomized Controlled Study
Brief Title: The Effects of Pilates on Posture and Physical Fitness Parameters in 5-6 Years Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Nazan Ozturk, PhD Lecturer, Physiotherapist, Aydin Adnan Menderes University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NOzturk
Record Dates: First submitted 2022-01-17; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Posture; Physical Fitness
Keywords: Pilates; Posture; Child; Physical Fitness; Preschool
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): The Pilates Group completed a 10-week. The intervention was performed in 20 sessions. The exercise program was created based on books and from the booklet acquired in the APPI Pilates Method training courses. Since the study was in preschool children, the basic level of Pilates was performed. Each exercise was performed 5 times for 30 minutes each twice a week .
  Interventions: Other: Pilates exercises
- Control (No Intervention): The Control Group did not perform any Pilates. The children in the CG continued their routine physical activities at school.

INTERVENTIONS:
Other: Pilates exercises — The Pilates Group completed a 10-week Pilates program. The intervention was performed in 20 sessions. In the first session, introduction and explanations regarding the principles and benefits of Pilates was made in a language that preschool children can understand. Exercises were supervised, and they were taught via gamification. In addition, the participation of the children was encouraged and stickers were given to increase their motivation at the end of the sessions. No adverse events occurred during intervention. The exercise program was created based on books and from the booklet acquired in the APPI Pilates Method training courses. Since the study was in preschool children, the basic level of Pilates was performed. Each exercise was performed 5 times for 30 minutes each twice a week.
  Arms: Pilates

SUMMARY:
The purpose of this non-randomized controlled study was to investigate the effects of Pilates on posture and physical fitness parameters in 5-6 years old healthy children.

As a result of this study, pilates can be applied as an alternative exercise that improves posture and physical fitness in children.

DETAILED DESCRIPTION:
The purpose of this non-randomized controlled study was to investigate the effects of Pilates on posture and physical fitness parameters in 5-6 years old healthy children.

As a result of this study, pilates can be applied as an alternative exercise that improves posture and physical fitness in children.

This study will answer whether pilates practice has an effect on posture and whether pilates has an effect on physical fitness parameters.Demographic information of the participants was recorded. Postural assessments were evaluated by the New York Posture Rating (NYPR) chart test and fitness was evaluated by the Eurofit test battery.

ELIGIBILITY:
Inclusion Criteria:

* Attending Aydın Bahçeşehir Kindergarten,
* Being allowed by her family to participate in the study
* Being a volunteer,
* Not having a diagnosed physical or mental illness that would prevent her from exercising.

Exclusion Criteria:

* Not being a volunteer,
* Having a health problem that prevents exercise.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
New York Posture Rating | immediately after application
  With this rating chart, postural changes that may occur in 13 different parts of the body are monitored and scored. The 13 body alignment segments include posterior views of the head, shoulders, spine, hip, feet, and arches, and lateral (left side) views of the neck, chest, shoulders, upper back, trunk, abdomen, and lower back. In this original version, each body segment was scored 5 (correct posture), 3 (slight deviation), or 1 (pronounced deviation). The total score obtained at the end of the test is maximum 65 and minimum 13
Eurofit test battery | immediately after application
  The Eurofit test battery is an easy to apply test battery for children to evaluate physical fitness. There are 9 tests within the Eurofit test battery to assess cardiorespiratory and motor fitness. These items are body balance, speed of arm movement, flexibility, handgrip strength, explosive force, abdominal muscle strength, shoulder muscles strength, running speed, and cardiovascular endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Bahcesehir Preschool, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk N, Unver F. The effects of pilates on posture and physical fitness parameters in 5-6 years old children: A non-randomized controlled study. J Bodyw Mov Ther. 2022 Jul;31:153-158. doi: 10.1016/j.jbmt.2022.03.009. Epub 2022 Mar 20. PMID 35710213